CLINICAL TRIAL: NCT04980118
Title: A Standardized Integral Nutritional Intervention 1 and Physical Activity Program
Brief Title: A Nutritional Intervention and Physical Activity Program Reduce Body Weight in Women Newly Diagnosed With Breast Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HULP 3114
Record Dates: First submitted 2019-09-12; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer; Body Weight Changes; Weight Loss; Nutrition Related Cancer
MeSH Terms: conditions — Breast Neoplasms; Body Weight Changes; Weight Loss | interventions — Control Groups; Nutritional Status

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Individual nutritional intervention.
  Interventions: Behavioral: Control group
- Experimental group (Experimental): Individual nutritional intervention with two groupal sessions and physical activity.
  Interventions: Behavioral: Nutrition and physical activity group

INTERVENTIONS:
Behavioral: Control group — A nutritional intervention program that consisted of two individual nutritional consults.
  Arms: Control group
Behavioral: Nutrition and physical activity group — A nutritional and physical activity intervention program that consisted of two individual nutritional consults and five nutritional group lectures.
  Arms: Experimental group

SUMMARY:
To evaluate a nutritional intervention for women newly diagnosed with breast cancer on a weight control and physical activity program.

DETAILED DESCRIPTION:
56 women newly diagnosed with breast cancer from the Department of Medical Oncology of La Paz University Hospital, Madrid, Spain.

A nutritional and physical activity intervention program that consisted of two individual nutritional consults and five nutritional group lectures was conducted by physicians of the Nutrition Unit during one year.

ELIGIBILITY:
Inclusion Criteria:

* Years: ≥18
* Sex: Female
* Newly diagnosed breast cáncer

Exclusion Criteria:

* Patients who have disseminated disease.
* Associated eating behavior disorders.
* Patients with dementia, mental illness or decreased cognitive function.
* Consumption of drugs or substances to lose weight (except in those cases in which it is suspended 15 days before starting the study).
* Presence of disease that may interfere with weight loss: severe psychiatric illness, uncontrolled hypothyroidism.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 56 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To evaluate a nutritional intervention for women newly diagnosed with breast cancer 9 weight control and physical activity program. | Six months
  To examine the frequency of food consumption

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gómez Candela, Msc, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Institute for Health Research IdiPAZ, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No